CLINICAL TRIAL: NCT02510040
Title: A Prospective Observational Study of Adult Strabismus
Acronym: SAS1
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SAS1; 2U10EY011751 (NIH)
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Convergence Insufficiency; Divergence Insufficiency; Hypertropia
Keywords: Convergence Insufficiency; Divergence Insufficiency; Small-angle Hypertropia; Strabismus
MeSH Terms: conditions — Ocular Motility Disorders; Strabismus | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Convergence insufficiency: Eligible adults with convergence insufficiency can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Interventions: Device: Prism; Other: Orthoptic Exercises; Procedure: Eye Muscle Surgery; Procedure: Botox Injection
- Divergence insufficiency: Eligible adults with divergence insufficiency can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Interventions: Device: Prism; Other: Orthoptic Exercises; Procedure: Eye Muscle Surgery; Procedure: Botox Injection
- Small-angle hypertropia: Eligible adults with small-angle hypertropia can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Interventions: Device: Prism; Other: Orthoptic Exercises; Procedure: Eye Muscle Surgery; Procedure: Botox Injection

INTERVENTIONS:
Device: Prism — Ground-in or Fresnel prism
Other: Orthoptic Exercises — Orthoptic exercises- fusion, convergence, divergence, and others, including computer-based therapy
Procedure: Eye Muscle Surgery — * Bilateral medial rectus muscle resection surgery
  * Single medial rectus muscle resection surgery
  * Recess lateral rectus muscle resection medial rectus muscle surgery
  * Bilateral lateral rectus muscle recession surgery
  * Single lateral rectus muscle recession surgery
  * Bilateral lateral rectus muscle resection surgery
  * Single lateral rectus muscle resection surgery
  * Recess medial rectus muscle resection lateral rectus muscle surgery
  * Bilateral medial rectus muscle recession surgery
  * Single medial rectus muscle recession surgery
  * Vertical rectus muscle recession surgery
  * Vertical rectus muscle mini-tenotomy (snip) surgery
Procedure: Botox Injection — Botulinum toxin injection
  Other Names: Botulinum toxin injection

SUMMARY:
The purpose of this study is to describe clinical characteristics, treatments, and one-year outcomes of adults with convergence insufficiency, divergence insufficiency, or small angle hypertropia.

DETAILED DESCRIPTION:
The purpose of this study is to describe clinical characteristics, treatments, and one-year outcomes of adults with convergence insufficiency, divergence insufficiency, or small angle hypertropia. Treatment comparisons within the studied conditions will also be done to help develop future studies.

ELIGIBILITY:
Eligibility Criteria for Convergence Insufficiency (CI) Group:

The following inclusion criteria must be met for the subject to be enrolled into the study:

* Adults ≥18 years of age (adult onset of CI not required)
* No strabismus surgery within the past 10 years
* CI Symptom Survey score ≥21 points
* Near exodeviation of ≥4∆ and at least 4∆ larger than at distance by PACT
* Distance exodeviation ≤15∆ by PACT
* Vertical deviation ≤2∆ at distance and near by PACT
* No constant exotropia at distance or near
* Reduced positive fusional vergence (PFV) at near (<20∆ or fails Sheard's criterion that the PFV measures less than twice the magnitude of the near phoria)
* Near point of convergence (NPC) of ≥6 cm break
* Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
* No paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* No monocular diplopia
* No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation.
* No inferior or superior oblique overaction defined as 2+ or greater
* Ability to fuse with prism in space (see section 2.4.1)
* Ability to understand and complete a survey
* Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
* If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment
* Single treatment modality is planned (e.g., no combined prism and orthoptic exercises)
* Treatment to be initiated has not been used within the past one year

Eligibility Criteria for Divergence Insufficiency (DI) Group:

The following inclusion criteria must be met for the subject to be enrolled into the study:

* Adults ≥18 years of age
* Adult-onset DI (at ≥18 years of age)
* No prior strabismus surgery
* Symptoms of diplopia at distance with a frequency of sometimes or worse in primary position (in current glasses if wearing glasses)
* Distance esodeviation of 2∆ to 30∆ and at least 50% larger than at near by PACT
* No more than 5∆ difference between right and left gaze by PACT
* No more than 10∆ difference between the primary position at distance and either upgaze or downgaze ≤10∆ by PACT
* Any coexisting vertical deviation must be less than distance esodeviation and ≤10∆ by PACT
* Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
* No paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* No monocular diplopia
* No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation
* No inferior or superior oblique overaction defined as 2+ or greater
* Ability to fuse with prism in space (see section 2.4.2)
* Ability to understand and complete a survey
* Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
* If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment
* Single treatment modality planned (e.g., no combined prism and orthoptic exercises)
* Treatment to be initiated has not been used within the past one year

Eligibility Criteria for Small-angle Hypertropia (HT) Group:

The following inclusion criteria must be met for the subject to be enrolled into the study:

* Adults ≥18 years of age
* Adult-onset HT (at ≥18 years of age)
* No prior strabismus surgery
* Symptoms of diplopia at distance or near with a frequency of sometimes or worse in primary or reading position (in current glasses if wearing glasses)
* Vertical deviation ≥1∆ to ≤10∆ at distance and near by PACT
* No more than 4∆ difference from the primary in any gaze position by PACT
* Any coexisting esodeviation must be less than the vertical deviation
* Any coexisting exodeviation ≤10∆ by PACT
* No convergence insufficiency as defined in section 2.2.1
* Visual acuity 20/50 or better in both eyes by ETDRS or Snellen
* No paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* No restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* No monocular diplopia
* No paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation.
* No inferior or superior oblique overaction defined as 2+ or greater
* Ability to fuse with prism in space (see section 2.4.3)
* Ability to understand and complete a survey
* Investigator is initiating treatment with prism, orthoptic exercises, botulinum toxin injection or surgery
* If initiating treatment with botulinum toxin or surgery, planned injection or surgery to be within 60 days of enrollment
* Single treatment modality planned (e.g., no combined prism and orthoptic exercises)
* Treatment to be initiated has not been used within the past one year

Exclusion Criteria for Convergence Insufficiency (CI) Group:

The following criteria exclude a subject from enrollment into the study:

* Strabismus surgery within the past 10 years
* CI Symptom Survey score ≥21 points
* Near exodeviation of ≤4∆ and at least 4∆ larger than at distance by PACT
* Distance exodeviation ≥15∆ by PACT
* Vertical deviation ≥2∆ at distance and near by PACT
* Constant exotropia at distance or near
* Near point of convergence (NPC) of ≤6 cm break
* Visual acuity worse than 20/50 either eye by ETDRS or Snellen
* Paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* Restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* Monocular diplopia
* Paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease. Patients with Parkinson's disease can be enrolled if non-paretic deviation.
* Inferior or superior oblique overaction defined as 2+ or greater
* Inability to fuse with prism in space (see section 2.4.1)
* Inability to understand and complete a survey
* Treatment to be initiated has already been used within the past one year

Exclusion Criteria for Divergence Insufficiency (DI) Group:

The following criteria exclude a subject from enrollment into the study:

* No adult-onset DI (at ≥18 years of age)
* Prior strabismus surgery
* Distance esodeviation outside the range of 2∆ to 30∆ and less than 50% larger than at near by PACT
* More than 5∆ difference between right and left gaze by PACT
* More than 10∆ difference between the primary position at distance
* Any coexisting vertical deviation more than distance esodeviation and ≥10∆ by PACT
* Visual acuity worse than 20/50 in either eye by ETDRS or Snellen
* Paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* Restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* Monocular diplopia
* Paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease.
* Inferior or superior oblique overaction defined as 2+ or greater
* Inability to fuse with prism in space (see section 2.4.2)
* Inability to understand and complete a survey
* Treatment to be initiated has already been used within the past one year

Exclusion Criteria for Small-angle Hypertropia (HT) Group:

The following criteria exclude a subject from enrollment into the study:

* No adult-onset HT (at ≥18 years of age)
* Prior strabismus surgery
* Vertical deviation ≤1∆ or ≥10∆ at distance and near by PACT
* More than 4∆ difference from the primary in any gaze position by PACT
* Coexisting esodeviation must not be less than the vertical deviation
* Coexisting exodeviation ≥10∆ by PACT
* Convergence insufficiency as defined in section 2.2.1
* Visual acuity worse than 20/50 in either eye by ETDRS or Snellen
* Paralytic strabismus (e.g., 3rd, 4th, or 6th cranial nerve palsies, skew deviation, Duane syndrome)
* Restrictive strabismus (e.g., blowout fracture, thyroid eye disease, post scleral buckle, Brown syndrome)
* Monocular diplopia
* Paretic strabismus, thyroid eye disease, myasthenia gravis, chronic progressive external ophthalmoplegia, or eye movement abnormalities associated with known neurological disease.
* Inferior or superior oblique overaction defined as 2+ or greater
* Inability to fuse with prism in space (see section 2.4.3)
* Inability to understand and complete a survey
* Treatment to be initiated has already been used within the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earl R Crouch, III, MD, Study Chair — Virginia Pediatric Eye Center
Locations (1):
- Earl R. Crouch, III, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the Pediatric Eye Disease Investigator Group (PEDIG) public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the protocol and publication of the primary manuscript, the data will be made available for the duration of the grant and any future grants.
Access Criteria: public

REFERENCES:
- [Result] Crouch ER, Dean TW, Kraker RT, Miller AM, Kraus CL, Gunton KB, Repka MX, Marsh JD, Del Monte MA, Luke PA, Peragallo JH, Lee KA, Wheeler MB, Daley TJ, Wallace DK, Cotter SA, Holmes JM; Pediatric Eye Disease Investigator Group. A prospective study of treatments for adult-onset divergence insufficiency-type esotropia. J AAPOS. 2021 Aug;25(4):203.e1-203.e11. doi: 10.1016/j.jaapos.2021.02.014. Epub 2021 Jul 13. PMID 34271207
- [Result] Lorenzana IJ, Leske DA, Hatt SR, Dean TW, Jenewein EC, Dagi LR, Beal CJ, Pang Y, Retnasothie DV, Esposito CA, Erzurum SA, Aldrich AE, Crouch ER, Li Z, Kraker RT, Holmes JM, Cotter SA; Pediatric Eye Disease Investigator Group; Pediatric Eye Disease Investigator Group. Relationships among Clinical Factors and Patient-reported Outcome Measures in Adults with Convergence Insufficiency. Optom Vis Sci. 2022 Sep 1;99(9):692-701. doi: 10.1097/OPX.0000000000001929. Epub 2022 Aug 2. PMID 35914096
- See also: PEDIG Public Website — http://pedig.jaeb.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Convergence Insufficiency: Eligible adults with convergence insufficiency can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Prism: Ground-in or Fresnel prism
  Orthoptic Exercises: Orthoptic exercises- fusion, convergence, divergence, and others, including computer-based therapy
  Eye Muscle Surgery: • Bilateral medial rectus muscle resection surgery
  * Single medial rectus muscle resection surgery
  * Recess lateral rectus muscle resection medial rectus muscle surgery
  * Bilateral lateral rectus muscle recession surgery
  * Single lateral rectus muscle recession surgery
  * Bilateral lateral rectus muscle resection surgery
  * Single lateral rectus muscle resection surgery
  * Recess medial rectus muscle resection lateral rectus muscle surgery
  * Bilateral medial rectus muscle recession surgery
  * Single medial rectus muscle recession surgery
  * Vertical rectus muscle recession surgery
  * Vertical rectus muscle mini-tenotomy (snip) surgery
  Botox Injection: Botulinum toxin injection
- Divergence Insufficiency: Eligible adults with divergence insufficiency can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Prism: Ground-in or Fresnel prism
  Orthoptic Exercises: Orthoptic exercises- fusion, convergence, divergence, and others, including computer-based therapy
  Eye Muscle Surgery: • Bilateral medial rectus muscle resection surgery
  * Single medial rectus muscle resection surgery
  * Recess lateral rectus muscle resection medial rectus muscle surgery
  * Bilateral lateral rectus muscle recession surgery
  * Single lateral rectus muscle recession surgery
  * Bilateral lateral rectus muscle resection surgery
  * Single lateral rectus muscle resection surgery
  * Recess medial rectus muscle resection lateral rectus muscle surgery
  * Bilateral medial rectus muscle recession surgery
  * Single medial rectus muscle recession surgery
  * Vertical rectus muscle recession surgery
  * Vertical rectus muscle mini-tenotomy (snip) surgery
  Botox Injection: Botulinum toxin injection
- Small-angle Hypertropia: Eligible adults with small-angle hypertropia can be treated with prism, orthoptic exercises, eye muscle surgery, or botox injection, per the investigator's usual clinical practice.
  Prism: Ground-in or Fresnel prism
  Orthoptic Exercises: Orthoptic exercises- fusion, convergence, divergence, and others, including computer-based therapy
  Eye Muscle Surgery: • Bilateral medial rectus muscle resection surgery
  * Single medial rectus muscle resection surgery
  * Recess lateral rectus muscle resection medial rectus muscle surgery
  * Bilateral lateral rectus muscle recession surgery
  * Single lateral rectus muscle recession surgery
  * Bilateral lateral rectus muscle resection surgery
  * Single lateral rectus muscle resection surgery
  * Recess medial rectus muscle resection lateral rectus muscle surgery
  * Bilateral medial rectus muscle recession surgery
  * Single medial rectus muscle recession surgery
  * Vertical rectus muscle recession surgery
  * Vertical rectus muscle mini-tenotomy (snip) surgery
  Botox Injection: Botulinum toxin injection
Period: Overall Study
Arm/Group | Convergence Insufficiency | Divergence Insufficiency | Small-angle Hypertropia
Started | 81 | 114 | 22
Completed | 63 | 111 | 21
Not Completed | 18 | 3 | 1
Not completed — Deemed no longer eligible | 18 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convergence Insufficiency | Divergence Insufficiency | Small-angle Hypertropia | Total
Number analyzed (Participants) | 63 | 111 | 21 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (18.6) | 67.4 (13.7) | 68.6 (13.0) | 59.5 (19.4)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38.2 [25.6 to 57.2] | 71.2 [60.8 to 75.7] | 71.5 [65.7 to 76.6] | 65.3 [44.2 to 74.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 74 | 10 | 132
  Male | 15 | 37 | 11 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 107 | 19 | 158
  Non-white | 31 | 4 | 2 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptom Success at 10 Weeks
Description: In the convergence insufficiency group, the primary outcome will be symptom success at the 10-week and 12-month visit, defined as improvement of CI Symptom Survey (CISS) score of at least 9 points and an outcome score of <21 points. In the divergence insufficiency group, the primary outcome will be symptom success at the 10-week and 12-month visit, defined as diplopia "rarely" or "never" in primary position at distance on the diplopia questionnaire. In the small-angle hypertropia group, the primary outcome will be symptom success at the 10-week and 12-month visit, defined as diplopia "rarely" or "never" both in primary position at distance and in reading position on the diplopia questionnaire.
Time Frame: 10 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Convergence Insufficiency | Divergence Insufficiency | Small-angle Hypertropia
Number analyzed (Participants) | 54 | 104 | 21
Participants | 25 | 91 | 12

2. Primary Outcome: Number of Participants With Symptom Success at 12 Months
Description: as for outcome 1
Time Frame: 12 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Convergence Insufficiency | Divergence Insufficiency | Small-angle Hypertropia
Number analyzed (Participants) | 54 | 98 | 18
Participants | 25 | 73 | 6

3. Secondary Outcome: Mean of Near Point of Convergence in Convergence Insufficiency Group
Description: Near point of convergence (convergence insufficiency group only).
Time Frame: 12 months after enrollment
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Convergence Insufficiency
Number analyzed (Participants) | 57
centimeters | 14.1 (6.2)

4. Secondary Outcome: Mean Positive Fusional Vergence in Convergence Insufficiency Group
Description: Positive fusional vergence (convergence insufficiency group only).
Time Frame: 12 months after enrollment
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Convergence Insufficiency
Number analyzed (Participants) | 57
prism diopters | 11.6 (7.1)

5. Secondary Outcome: Adult Strabismus 20 Questionnaire Score (DI)
Description: Adult Strabismus Quality of Life Questionnaire (AS-20) For AS-20, scores are reported for the following subscales. A total score will not be reported.
  1. Self-perception score
  2. Interaction score
  3. Reading function score
  4. General function score Values for each subscale range from 0 to 100. 0 indicates poor quality of life (the patient reported "always" for all questions) and 100 represents good quality or life (patient reported "never" for all questions)
Time Frame: 12 months after enrollment
Population: This information was only collected and analyzed for the DI and CI arms. The HT arm cannot be reported since it was not collected. The CI arm data is currently being analyzed, and will be added to the record when analysis is complete, results are expected May 2021.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Divergence Insufficiency
Number analyzed (Participants) | 111
score on a scale
  General Function Score | 62 (22)
  Reading Function Score | 71 (23)
  Self Perception Score | 87 (19)
  Interaction Score | 94 (11)

6. Secondary Outcome: Mean Convergence Insufficiency Symptom Survey Score
Description: Mean Convergence Insufficiency Symptom Survey Score (convergence insufficiency group only) For CISS, the range is from 0 (having no symptoms of CI) to 60 (always showing all symptoms of CI).
Time Frame: 12 months after enrollment
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Convergence Insufficiency
Number analyzed (Participants) | 57
points | 37.5 (9.1)

7. Secondary Outcome: Adult Strabismus 20 Questionnaire Score (CI)
Description: Adult Strabismus Quality of Life Questionnaire (AS-20) For AS-20, scores are reported for the following subscales. A total score will not be reported.
  Self-perception score Interaction score Reading function score General function score Values for each subscale range from 0 to 100. 0 indicates poor quality of life (the patient reported "always" for all questions) and 100 represents good quality or life (patient reported "never" for all questions)
Time Frame: 12 months after enrollment
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Convergence Insufficiency
Number analyzed (Participants) | 57
points
  General Function | 55.7 (24.6)
  Reading Function | 43.9 (22.2)
  Interaction | 92.2 (14.7)
  Self Perception | 83.8 (22.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected since treatment was prescribed per usual standard of care.
Description: Per the study protocol (sections 4.4.1 and 4.5)
  Risks of Examination Procedures The procedures in this study are part of daily eye care practice in the United States and pose no known risks.
  Reporting of Adverse Events No treatments are being prescribed that are not part of usual care. Investigators will abide by local IRB reporting requirements.
Arm/Group | Convergence Insufficiency | Divergence Insufficiency | Small-angle Hypertropia
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT02510040/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT02510040/SAP_002.pdf
  • Informed Consent Form (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT02510040/ICF_001.pdf